CLINICAL TRIAL: NCT07153211
Title: Analysis of Selected Biochemical Parameters in Cerebrospinal Fluid and Peripheral Blood in the Treatment of Neuropathic Pain Using Spinal Cord Stimulation (SCS) Assessment of the Mechanism of Action of SCS and the Potential of Biochemical Studies in Therapy Planning and Monitoring
Brief Title: Analysis of Selected Biochemical Parameters in Cerebrospinal Fluid and Peripheral Blood in the Treatment of Neuropathic Pain Using Spinal Cord Stimulation (SCS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pawel Sokal (Other)
Collaborators: Department of Neurosurgery Collegium Medicum Nicolaus Copernicus University (Unknown); Nicolaus Copernicus University in Toruń, Collegium Medicum in Bydgoszcz (Other)
Responsible Party: Sponsor-Investigator, Pawel Sokal, Professor, Jan Biziel University Hospital No 2 in Bydgoszcz
Organization: Jan Biziel University Hospital No 2 in Bydgoszcz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KB345/2022
Record Dates: First submitted 2025-08-10; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Neuropathic Pain; Chronic Pain; Spinal Cord Stimulation (SCS)
Keywords: spinal cord stimulation; neuropathic pain; immunomodulatory effects of scs
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with SCS - tonic stimulation (Experimental): We plan to include 30-50 patients with PSPS or CRPS undergoing SCS implantation. Blood will be collected before surgery and 2-3 weeks after; CSF during both procedures. Pain (VAS), disability (ODI), neurological status, muscle tone, and analgesic intake will be assessed. Temporary stimulation will last 2-3 weeks before IPG implantation or electrode removal. Samples will be processed and analyzed via ELISA in our Biochemistry Department using established protocols.
  Interventions: Diagnostic Test: Immunological Factors

INTERVENTIONS:
Diagnostic Test: Immunological Factors — Assessment of interleukins and other molecues in CSF and blood of patients with SCS.

SUMMARY:
This project aims to identify key cells and molecules involved in the development and modulation of neuropathic pain treated with spinal cord stimulation (SCS). By measuring concentrations of selected inflammatory mediators and signaling molecules (e.g., IL-1β, IL-6, IL-17, IL-33, BDNF, VEGF, GABA) in the blood and cerebrospinal fluid (CSF) of patients undergoing SCS, the study seeks to better understand the mechanism of action of SCS. The findings may allow the development of predictive biomarkers, help tailor stimulation parameters, and support complementary pharmacotherapy. The project also explores differences in response to various stimulation types and the role of glial cells in SCS efficacy, with a view to improving patient outcomes through more personalized neuromodulation strategies.

DETAILED DESCRIPTION:
1. The Aim of the Project

   The aim of this project is to measure the concentrations of selected inflammatory mediators and other signalling molecules in the blood and cerebrospinal fluid (CSF) of patients undergoing spinal cord stimulation (SCS). The goal is to identify which cells and molecules are crucial in the development of neuropathic pain and its treatment via SCS. This will provide insight into the mechanisms underlying SCS and enhance our understanding of how it works.

   Additionally, the correlation between the concentrations of these molecules and patients' clinical status, treatment outcomes (whether successful or not), and especially blood concentrations of certain markers, may allow for the development of simple tools for predicting the response to a particular type of stimulation, monitoring treatment effectiveness, and identifying potential complementary pharmacotherapies.

   Previous research conducted by my team, which forms the basis for this project, has shown that SCS affects iron and calcium metabolism and that different types of stimulation vary in their effectiveness in reducing pain. This variation may stem from the superiority of one method over another or from patient-specific factors, which this study aims to clarify.
2. Importance of the Project

   SCS has been successfully used to treat neuropathic pain for over fifty years. Despite ongoing advancements-such as new devices and stimulation techniques-the exact mechanism of SCS remains unknown. Not only is it unclear which cells mediate pain signal inhibition, but even the precise target site of stimulation is still under debate. Genomic studies on animal models have so far failed to resolve this issue.

   Recent theories suggest that stimulation of interneurons in the posterior horns of the spinal cord inhibits sensory neurons. However, given that the glial-to-neuron ratio in the spinal cord (where electrodes are typically placed) is around 20:1, it seems unlikely that glial cells play only a passive role. Many types of glial cells are involved in neurotransmitter transport and processing, mediate inflammatory responses, and can be depolarized themselves. Thus, the mechanisms of neuropathic pain and its modulation by SCS may be more complex and heterogeneous than initially assumed. This complexity may explain why some patients respond poorly to SCS or respond better to certain stimulation types, even when their clinical and radiological conditions appear similar to those of patients who experience significant pain relief.
3. Concept and General Research Plan

   Inflammation is a universal response to injury, infection, or other disturbances and involves immune system activation and changes in the function, phenotype, and number of local cells. It is, therefore, unsurprising that neuropathic pain is associated with inflammation in the nervous system, including the spinal cord.

   To assess this, the project will measure levels of pro- and anti-inflammatory factors, as well as other molecules potentially linked to the inflammatory response at baseline and after 14 days of trial stimulation. Special attention will be given to the dynamic changes in these molecules following SCS. The following substances will be measured in CSF and serum:

   IL-1β, IL-4, IL-6, IL-10, IL-17, IL-33, VEGF, BDNF, GABA

   Animal studies have shown:

   IL-1β affects neuronal metabolism and depolarization and is involved in neuropathic pain mechanisms. SCS reduces IL-1β levels in damaged spinal cords.

   IL-6, stimulated partly by IL-1β, reduces pain intensity and enhances opioid sensitivity in rats.

   IL-17, produced by astrocytes, blocks neuronal inhibition and causes mechanical allodynia in healthy mice.

   IL-33, produced mainly by oligodendrocytes in the CNS, plays a key role in neuropathic pain pathogenesis.

   Progesterone and estradiol have neuroprotective effects, partly through reducing inflammation, which could influence individual variability in pain perception and SCS responsiveness.

   Other molecules under investigation are associated with inflammation or serve as trophic factors. They may participate in the pathomechanism of neuropathic pain, play a role in SCS treatment, or serve as clinically useful biomarkers. SCS has been associated with detectable changes in the production of certain interleukins. Some interleukins, such as IL-33, IL-6, and IL-1β, promote the expression of anti-apoptotic factors and support neuronal and glial cell survival via pathways like nuclear factor κB (NFκB). Importantly, changes in interleukin expression in neural tissue have been shown to correlate with changes in CSF concentrations.

   Despite promising animal model data, there is a significant lack of equivalent human studies. This project aims to address that gap. Changes in specific interleukin levels may help identify which glial cells respond to SCS and which molecules are key to the treatment's efficacy.
4. Materials and Methods

In the SCS procedure, two electrodes are placed on the dura mater, typically between the Th8-Th10 vertebrae. Patients undergo trial stimulation for 2-3 weeks. If effective, a second surgery is performed to implant a permanent pulse generator (IPG) under the skin in the lumbar region. This IPG can stimulate the spinal cord for up to 10 years, blocking pain signals.

Importantly, all patients included in this study would undergo these surgeries regardless of the research. The study involves only the collection of blood and CSF samples, along with additional monitoring and assessment. If the sample size permits, patients may be randomized into groups with different stimulation parameters, as described below.

We plan to include 20-50 patients with post-surgical pain syndrome (PSPS) and complex regional pain syndrome (CRPS) admitted for SCS implantation. Blood samples will be collected the day before or on the day of the first surgery, and again 2-3 weeks later. CSF samples will be collected during both the first and second procedures. Pain will be assessed using the VAS scale, and quality of life using the Oswestry Disability Index (ODI) questionnaire, completed preoperatively and again 2-3 weeks postoperatively. Patients will also keep a log of their pain medication use during the study. Neurological examinations, including assessments of deficits and muscle tone, will be performed preoperatively.

Initially, patients receive a temporary IPG for 2-3 weeks with standard tonic stimulation. If they respond well, a second surgery is performed for permanent IPG implantation. If not, alternative stimulation parameters may be tried, or electrodes may be removed upon the patient's request. Blood and CSF samples may be collected from both responders and non-responders during the second procedure.

If we include more than 40 patients, we aim to form subgroups based on stimulation parameters:

Tonic stimulation group

Burst stimulation (or equivalent) group

Sham group (pending bioethics committee approval)

Patients in the sham group will have electrodes implanted but will receive no stimulation during the trial period. After sample collection, proper stimulation will commence.

Samples will be immediately transported to the Department of Biochemistry at our university, where trained staff will process, freeze, and analyze them using ELISA kits. This method was developed during our previous studies.

After the final sample collection, stimulation parameters will be tailored individually for each patient based on their preferences and pain relief outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* PSPS or CRPS
* Neuropathic pain for at least 6 months

Exclusion Criteria:

* Drug/alcohol addiction
* Malignant tumour
* Psychiatric disorders
* Active infection
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | baseline and after 14 days of trial stimulation
  Oswestry Disability Index before and after trial stimulation
Pain reduction | baseline and after 14 days of trial stimulation
  VAS

SECONDARY OUTCOMES:
Changes in blood and CSF inflammatory markers | baseline and after 14 days of trial stimulation
  Changes in blood and CSF inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- Jan Bizel University Hospital, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No
No patient consent.